CLINICAL TRIAL: NCT07354152
Title: COmparison of the Use of a PERforator Flap Versus Total Skin GRAft in the Management of Loss of Substance After Resection of Cutaneous Melanoma - Pilot Study
Acronym: COPERGRAM1
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_UL_02
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stage II Cutaneous Melanoma
Keywords: melanoma; skin graft; perforator flap
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- skin graft (routine care): Skin grafting decided by the multidisciplinary tumor board
- perforator flap (routine care): perforator flap decided by the multidisciplinary tumor board

SUMMARY:
Melanoma is an aggressive and potentially fatal skin cancer and was the fifth most commonly diagnosed cancer among both men and women in the United States in 2022. When detected early, cutaneous melanoma has a favorable prognosis, with a 5-year survival rate exceeding 90%. Because melanoma frequently affects younger patients, wide local excision according to international guidelines may result in substantial functional and aesthetic morbidity.

Reconstruction is therefore a critical component of locoregional management and should aim to optimize functional and aesthetic outcomes without compromising oncologic control. To date, no consensus exists regarding the optimal reconstructive strategy. Skin grafts are often favored for their presumed ability to facilitate early detection of local recurrence but are associated with donor-site morbidity and suboptimal morphofunctional outcomes. Flap reconstruction has been reported to improve healing time and aesthetic results; however, it is not commonly considered first-line after melanoma excision, largely due to the unsubstantiated concern that flaps may delay recurrence detection. Notably, objective data supporting this concern are lacking.

Only two retrospective studies have addressed this issue. The largest, including 165 patients, reported that perforator-based pedicled flaps achieved favorable functional and aesthetic outcomes without adversely affecting locoregional disease control. A smaller study of facial melanoma similarly found immediate reconstruction with a facial artery perforator flap to be safe and aesthetically satisfactory.

In our institution, both skin grafts and flap reconstructions are used following multidisciplinary discussion. We therefore aim to comparatively evaluate wound healing after margin re-excision and patient-reported quality of life following melanoma excision, regardless of tumor stage or location, to determine whether one reconstructive approach provides superior clinical or functional benefit in routine practice.

DETAILED DESCRIPTION:
This study compares two groups of patients who underwent different standard-of-care reconstructive techniques following margin re-excision for stage II cutaneous melanoma, with the reconstructive approach selected during a multidisciplinary tumor board dedicated to melanoma management.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (≥ 18 years)
* Patients with cutaneous melanoma of any stage (I, II, or III) according to the AJCC Cancer Staging Manual, 8th edition (2017), diagnosed prior to surgery
* Non-closable surgical defect after margin re-excision

Exclusion Criteria:

* Patients with microscopic or macroscopic nodal involvement when the sentinel lymph node has been removed
* Patients with distant metastases identified on ultrasound and/or CT scan and/or PET-CT, when performed
* Surgical contraindication to perforator flap reconstruction
* Pregnant or breastfeeding women
* Patients without health insurance coverage
* Vulnerable individuals: persons deprived of liberty, under legal guardianship, or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for cutaneous melanoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
wound healing | up to 3 months
  To compare wound healing time, measured in days, between two groups of patients with stage II cutaneous melanoma of the trunk, abdomen, or limbs who underwent different reconstructive techniques following margin re-excision: skin grafting (gold standard) versus perforator-based flap reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Gaudian, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Study protocol + article
Supporting Information: Study Protocol